CLINICAL TRIAL: NCT00296257
Title: A Phase 2, Multi-Centre, Randomised, Double Blind, Placebo Controlled Study Evaluating the Efficacy, Safety and Pharmacokinetics of Two Doses of a Candidate Disease Modifying Anti-Rheumatic Drug (DMARD), (SMP-114 120 mg and 240 mg Once Daily), Administered in Combination With Ongoing Methotrexate Treatment in Patients With Active Rheumatoid Arthritis.
Brief Title: Assessment of Safety, Pharmacokinetics and Efficacy in a Combination Treatment With SMP-114
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Dainippon Sumitomo Pharma Europe LTd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2450174
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — rimacalib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SMP-114

SUMMARY:
To compare the efficacy of SMP-114 (120 and 240 mg/d) versus placebo in terms of the percentage of patients meeting the American College of Rheumatology criteria for 20% improvement in RA (ACR20) at week 24. The study hypothesis would be to demonstrate that the use of methotrexate and SMP-114 is more efficacious than Methotrexate alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged at least 18 years, with RA for a minimum of 6 months
* Has been receiving methotrexate treatment (stable for 8 weeks)
* Has active disease classified as ACR functional class of I, II or III

Exclusion Criteria:

* Has previously discontinued DMARD therapy due to hepatic intolerance
* Has received any DMARD in addition to methotrexate during the 4 weeks prior to randomisation
* Is receiving more than 2 DMARDs in addition to methotrexate at the time of screening
* Is receiving or has received Gold, leflunomide or biological agents including TNF/IL-1 inhibitors within the 8 weeks prior to randomisation
* Has previously failed 2 or more DMARDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2006-02; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of SMP-114 versus placebo in terms of the percentage of patients meeting the ACR criteria for 20% improvement in RA (ACR20) at Week 24.

SECONDARY OUTCOMES:
To compare efficacy of SMP-114 versus placebo after 24 weeks in terms of ACR50, ACR70, DAS28 and EULAR response.
To compare the efficacy of SMP-114 versus placebo in terms of change in core variables, time to response, Quality of Life, radiological measurements of joint damage, assessment of safety and tolerability, and PK measurements

CONTACTS AND LOCATIONS:
Overall Officials: David Scott, MD, FRCP, Principal Investigator — Kings College Hospital
Locations (42):
- Czechia (8):
  - Česká Lípa
  - České Budějovice
  - Hlučín
  - Ostrava Trebovice
  - Prague
  - Terezín
  - Uherské Hradiště
  - Zlín
- Germany (6):
  - Bad Nauheim
  - Freiburg im Breisgau
  - Hildesheim
  - Leipzig
  - Ratingen
  - Zerbst
- Hungary (8):
  - Békéscsaba
  - Budapest
  - Debrecen
  - Esztergom
  - Kecskemét
  - Komárom
  - Miskolc
  - Szombathely
- Netherlands (3):
  - Groningen
  - JD Alkmaar
  - Rotterdam
- Poland (8):
  - Częstochowa
  - Elblag
  - Katowice
  - Lublin
  - Sopot
  - Swietokrzyce
  - Szczecin
  - Warsaw
- United Kingdom (9):
  - Birmingham
  - Colchester
  - Greenock
  - Huddersfield
  - London
  - Maidstone
  - Metropolitan Borough of Wirral
  - Middlesbrough
  - Newcastle Upon Tyne and Wear